CLINICAL TRIAL: NCT07266571
Title: Pycnogenol (French Maritime Pine Bark) for the Treatment of Gulf War Illness
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Jarred Younger, Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 30015456; UAB (Other: UAB)
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Gulf War Syndrome
Keywords: Gulf War Illness; Pycnogenol; Botanical; French Maritime Pine Bark
MeSH Terms: conditions — Persian Gulf Syndrome | interventions — microcrystalline cellulose; pycnogenols

STUDY DESIGN:
Masking Description: This study is single-blind, participants will not know when they received placebo or pycnogenol. There are also four possible dosages for pycnogenol. Participants will also receive placebo (capsules with an inactive substance) at some point during the treatment phase of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants Receiving Botanicals (Experimental): Participants Receiving Botanicals
  Interventions: Other: Placebo; Dietary Supplement: Pycnogenol, 100mg; Dietary Supplement: Pycnogenol, 200mg; Dietary Supplement: Pycnogenol, 400mg; Dietary Supplement: Pycnogenol, 600mg

INTERVENTIONS:
Other: Placebo — The placebo being used in this study is microcrystalline cellulose. This will be taken orally, up to twice per day.
  Other Names: Microcrystalline Cellulose
Dietary Supplement: Pycnogenol, 100mg — Pycnogenol being used in this study is a commercially available dietary supplement and is classified as food by the FDA instead of a drug. This will be taken orally, up to twice per day.
  Other Names: French Maritime Pine Bark
Dietary Supplement: Pycnogenol, 200mg — Pycnogenol being used in this study is a commercially available dietary supplement and is classified as food by the FDA instead of a drug. This will be taken orally, up to twice per day.
  Other Names: French Maritime Pine Bark
Dietary Supplement: Pycnogenol, 400mg — Pycnogenol being used in this study is a commercially available dietary supplement and is classified as food by the FDA instead of a drug. This will be taken orally, up to twice per day.
  Other Names: French Maritime Pine Bark
Dietary Supplement: Pycnogenol, 600mg — Pycnogenol being used in this study is a commercially available dietary supplement and is classified as food by the FDA instead of a drug. This will be taken orally, up to twice per day.
  Other Names: French Maritime Pine Bark

SUMMARY:
The purpose of this research study is to determine how pycnogenol may reduce Gulf War Illness (GWI) symptom severity. The study will also examine the safety of this treatment and determine the optimal dosage. We believe that GWI involves inflammation in the body and brain that causes fatigue, pain, cognitive disruption, and other symptoms. Botanicals that reduce inflammation may help treat GWI.

DETAILED DESCRIPTION:
This study uses a decentralized design where individuals can participate from anywhere in the United States. Botanicals will be received by mail. Participants will also receive placebo (capsules with an inactive substance) during the treatment phase of the study. All participants will have been present in the Persian Gulf between 1990 and August 1991. This study will be tested on GWI participants recruited nationwide, with a total of 20 participants enrolled for the entire study. Participation will last 12 months.

The first stage of the study is the baseline phase. During this time, participants will complete weekly questionnaires about symptom severity ratings but will not take any capsules. The baseline stage will last for 30 days.

After the 30-day baseline, the treatment stage will begin. Capsules will be taken once in the morning, and once before bed. This study is single-blind, meaning that participants will not know when placebo or pycnogenol are received. There are also four possible dosages for pycnogenol.

The capsules will be packaged to indicate the order in which they should be taken. The capsules will be packaged in blister packs and shipped to participants. The capsules are designed to look the same throughout the study, though the contents can change. This treatment stage is the longest, lasting 10 months.

During the treatment stage, participants will also be asked to complete weekly questionnaires about GWI symptoms. These weekly questionnaires will also ask about changes in symptoms and overall quality of life, as well as changes in physical and mental health. Questionnaires can be completed on a smartphone, computer, or tablet. If participants do not have an appropriate device, or do not want to use your personal device, a tablet can be sent for the study. A research team member will speak with participants to set up electronic device connections and will verify the information is received.

At the end of the treatment stage, participants will stop taking capsules and will complete the end line stage. This stage is the same as the baseline stage in which participants will complete weekly symptom measures without taking capsules. This stage will last for 30 days.

After completion of the study, participants will be told when placebo was received, and what dosage(s) of treatment were received. Participants will also be shown how GWI severity changes over time.

While this study is long, it is designed to not be a significant burden to daily life. On most days, participation (taking morning capsules, taking evening capsules, and completing weekly symptom severity reports) should take approximately 2 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Meet the Kansas GWI case definition
* Meet the CDC GWI case definition
* Able to commit to a 12-month study
* Participants will be individuals in our Gulf War database who have already completed our other botanical trial, Curcumin, Resveratrol, and Stinging Nettle as Treatments for Gulf War Illness (NCT05377242).

Exclusion Criteria:

* Currently involved in another experimental treatment study
* Currently pregnant
* Have a blood clotting disorder
* Reported diagnosis of diabetes with a A1C greater than 9
* Use of contraindicated medications (see below):
* Anticoagulants (such as warfarin, heparin, etc.)
* Lithium
* Tacrolimus (Prograf)
* Cancer medications (Alkylating agents, antitumor antibiotics, Topoisomerase I inhibitors, Tamoxifen)
* Daily Use of Antiplatelet agents (e.g. aspirin, clopidogrel)
* Nitroglycerin
* Hypotension
* Need for surgery during study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in Physical Functioning Score of the VR-12 | 12 months
  This change will be measured using weekly surveys (ADD THE ACTUAL SCALE)
Change in Mental Functioning Score of the VR-12 | 12 months
  This change will be measured using weekly surveys (ADD THE ACTUAL SCALE)

CONTACTS AND LOCATIONS:
Overall Officials: Jarred Younger, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No